CLINICAL TRIAL: NCT04028505
Title: Terlipressin Bolus Versus Continuous Infusion in Patients With Variceal Hemorrhage
Brief Title: Terlipressin Infusion in Variceal Hemorrhage
Acronym: TT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, SHAHAB ABID, Professor and Head Section of Gastroenterology, Department of Medicine, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5209-Med-ERC-18
Record Dates: First submitted 2018-05-10; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Terlipressin Adverse Reaction
Keywords: Terlipressin Drug; Continuous Infusion; Bolus Form

STUDY DESIGN:
Intervention Model Description: Experimental Arm: Standard of care being given at AKUH + Continuous infusion of Terlipressin at a rate of 0.5mg/hour for the first 24 hours Comparator Arm: Standard of care being given at AKUH + Bolus infusion of Terlipressin at a frequency of 2mg every six hourly for first 24 hours
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Terlipressin Continuous Infusion (Experimental): Standard of care being given at AKUH + Continuous infusion of Terlipressin (Terlipressin Injectable Product) at a rate of 0.5mg/hour for the first 24 hours
  Interventions: Drug: Terlipressin Injectable Product
- Terlipressin Bolus Infusion (Active Comparator): Standard of care being given at AKUH + Bolus infusion of Terlipressin (Terlipressin Injectable Product) at a frequency of 2mg every six hourly for first 24 hours
  Interventions: Drug: Terlipressin Injectable Product

INTERVENTIONS:
Drug: Terlipressin Injectable Product — Intravenous terlipressin will be obtained from Clinical Trials Unit, AKUH pharmacy in standard IV infusion form.
  Participants who are randomized to the intervention arm will be administered a continuous infusion of Terlipressin at a rate of 0.5mg/hour for the first 24 hours. Participants randomized into the control group will be administered a bolus form of Terlipressin at a rate of 2mg every six hourly for the first 24 hours respectively. In case of weekends/public holidays intravenous terlipressin will be obtained from the main pharmacy of AKUH.
  Other Names: Novapressin

SUMMARY:
Randomized, open label study of intravenous terlipressin infusion vs. bolus for the treatment of variceal hemorrhage. 24 hour regimen consisting of intravenous terlipressin will be used either at a rate of 0.5mg/hour or 2mg bolus every 4 hourly. Participants will be randomized into intervention and control arm using block randomization by computer generated random numbers. Efficacy will be assessed by clinical improvement in symptoms and signs of GI bleed. To assess safety, frequency and degree of adverse reactions will be observed. Periodic assessments until 5 days will be done consisting of physical examination, safety assessments, vital signs and lab tests.

DETAILED DESCRIPTION:
Randomized, open label trial, conducted on patients admitted with acute variceal hemorrhage at The Aga Khan University Hospital, Karachi (AKUH). Patients will be followed in clinic after discharge to assess survival for 6 weeks.

Intravenous terlipressin will be obtained from Clinical Trials Unit, AKUH pharmacy in standard IV infusion form. Following complete clinical and laboratory evaluation, assessing the patient for eligibility, informed consent will be obtained from all the participants who are willing to be part of this study. After obtaining the informed consent, study participants will be randomized into the intervention arm (continuous infusion of Terlipressin) or the control arm (bolus form of Terlipressin). Participants who are randomized to the intervention arm will be administered a continuous infusion of Terlipressin at a rate of 0.5mg/hour for the first 24 hours. Participants randomized into the control group will be administered a bolus form of Terlipressin at a rate of 2mg every six hourly for the first 24 hours respectively. In case of weekends/public holidays intravenous terlipressin will be obtained from the main pharmacy of AKUH.

The trial will be conducted in in-patient units of AKUH where eligible patients are admitted. It may include emergency room, special care unit and general ward. Moreover, patients will be followed up by phone calls and in outpatient's clinics to assess survival six weeks post discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 60 years
2. Either gender
3. A diagnosis of liver cirrhosis;
4. Initial presentation with acute gastroesophageal variceal bleeding
5. Willing to provide informed consent to participate in the study (by study subject or next of kin)

Exclusion Criteria:

1. Age < 18 or > 60 years
2. Not willing to provide consent due to any reason
3. No liver cirrhosis
4. Acute upper gastrointestinal bleeding unrelated to varices;
5. Use of somatostatin or octreotide.
6. Hepatocellular Carcinoma (HCC)outside Milan's criteria
7. Advance cardiovascular, pulmonary or renal disease (e.g. asthma, hypertension, arrhythmia, renal insufficiency)
8. History of hypersensitivity to Terlipressin
9. Pregnancy
10. Patients already admitted at AKUH who develop upper GI bleed during admission.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-04-25 (Estimated); Study Completion 2020-10-25 (Estimated)

PRIMARY OUTCOMES:
Reduction in tachycardia, measured through heart rate (>100 bpm) being displayed in the electronic monitors in wards, emergency room and out-patient clinics | 6 weeks (Overall length of follow-up)
  It will be assessed by trained research coordinator as; the number of study participants with 20% reduction in tachycardia as compared to the baseline between the two arms.
Improvement in mean arterial pressure, being displayed in the electronic monitors in wards, emergency room and out-patient clinics | 6 weeks (Overall length of follow-up)
  It will be assessed by trained research coordinator as; the number of study participants with 20% improvement in mean arterial pressure as compared to the baseline between the two arms.
  Adverse events related to terlipressin, such as hyponatremia, diarrhea, abdominal pain; arterial hypertension should be reported to the primary gastroenterologist between the two arms.
In-patient hospital mortality, assessed through medical records. | Admission of patient till death in the hospital
  It will be assessed through medical records, by a trained research coordinator as the number of study participants dying within the hospital between the two arms.
Failure to control bleeding as assessed by physiological parameters in the blood | Admission of patient till discharge from the hospital
  It will be assessed by a trained research coordinator as the number of participants having fresh hematemesis and 3 gm drop in hemoglobin (9% drop in hematocrit) within a 24 hours' time period between the two arms.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 6 weeks (Overall length of follow-up)
  It will be assessed by trained research coordinator as; the number of participants having experienced any adverse events such as hyponatremia, diarrhea, abdominal pain, arterial hypertension, 5 days after having terlipressin drug, between the two arms.

SECONDARY OUTCOMES:
Out of hospital mortality assessed through telephonic interviews from patient's caregiver | 5 weeks after being discharged from the hospital
  It will be assessed by trained research coordinator as; the number of participants dying after being discharged from the hospital between the two arms within the follow-up time period of the study.
Failure to control bleeding as assessed by physiological parameters in the blood | 5 weeks after being discharged from the hospital
  It will be assessed by trained research coordinator as the number of participants having fresh hematemesis and 3 gm drop in hemoglobin (9% drop in hematocrit) after being discharged from the hospital till three subsequent follow-up visits between the two arms.
Prolong hospital stay (> 5 days) as assessed through medical records and pre-designed questionnaire | 5 days after admission till being discharged from the hospital
  It will be assessed by trained research coordinator as; the number of participants having stayed in the hospital for more than five days between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Shahab Abid, PhD,FRCP, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No